CLINICAL TRIAL: NCT04845880
Title: Evaluation of IgG Neutralizing Antibodies to SARS-CoV-2 Among Healthcare Workers Who Frequently Encountered COVID-19 Patients in Our Hospital
Brief Title: SARS Cov_2 Incidence of Healthy Health Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Hikmet Eda Aliskan (Unknown); Hatice Hale Gumus (Unknown); Ilker Odemis (Unknown); Zuhal Ekici Unsal (Unknown)
Responsible Party: Principal Investigator, Hasan Yesilagac, Specialist Doctor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: KA20/449
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: SARS COV-2 IgG Levels on Health Workers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS Cov_2 Incidence of Healthy Health Workers (Other)
  Interventions: Diagnostic Test: Spike protein (S) or the nucleocapsid (N) of SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Spike protein (S) or the nucleocapsid (N) of SARS-CoV-2 — Blood level of spike protein (S) or the nucleocapsid (N) of SARS-CoV-2

SUMMARY:
Since the severe acute respiratory syndrome Coronavirus-2 (SARS-CoV-2) first emerged in Wuhan, China, on 12 December 2019, it has spread rapidly across the world and developed into a pandemic. The pandemic has affected over 100 countries and regions, with over 132 million confirmed cases of COVID-19. The rapid spread of SARS-CoV-2 has caused considerable harm to public health and the economy. Alongside other laboratory tests and clinical findings of the COVID-19 infection, serological testing may be beneficial for epidemiological monitoring and outbreak control. The determination of antibodies enables confirmation of the SARS-CoV-2 infection in asymptomatic patients in addition to those with typical symptoms. In this study, we aimed to determine the SARS-CoV-2 seroprevalence and the IgG antibody levels among healthcare workers who frequently encountered COVID-19 patients in our hospital.

ELIGIBILITY:
Inclusion Criteria:

Healthy Health Workers - SARS COV-2 PCR (-)

Exclusion Criteria:

Health Workers - SARS COV-2 PCR (+) Pregnancy Autoimmune diseases Received immunosuppressive therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of IgG Neutralizing Antibodies to SARS-CoV-2 Among Healthcare Workers Who Frequently Encountered COVID-19 patients in Our Hospital | 6 months
  Determining antibody levels and seroprevalence of healthy healthcare workers

CONTACTS AND LOCATIONS:
Locations (1):
- Adana Dr. Turgut Noyan Application and Research Center, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Yang W, Cao Q, Qin L, Wang X, Cheng Z, Pan A, Dai J, Sun Q, Zhao F, Qu J, Yan F. Clinical characteristics and imaging manifestations of the 2019 novel coronavirus disease (COVID-19):A multi-center study in Wenzhou city, Zhejiang, China. J Infect. 2020 Apr;80(4):388-393. doi: 10.1016/j.jinf.2020.02.016. Epub 2020 Feb 26. PMID 32112884
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261